CLINICAL TRIAL: NCT02339376
Title: Treating Deep Seizure Foci With Noninvasive Surface Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Bernard Chang, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014P000216
Record Dates: First submitted 2015-01-08; First posted 2015-01-15 (Estimated); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy, Temporal Lobe
MeSH Terms: conditions — Epilepsy, Temporal Lobe | interventions — Neuronavigation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Group 1 (Experimental): Low-frequency repetitive transcranial magnetic stimulation: 30-minute sessions of 1-Hz continuous stimulation at 95% resting motor threshold, with one session each day over 10 consecutive weekdays
  Interventions: Device: Low-frequency repetitive transcranial magnetic stimulation
- Group 2 (Experimental): High-frequency repetitive transcranial magnetic stimulation: 30-minute sessions of 10-Hz continuous stimulation at 110% resting motor threshold, with one session each day over 10 consecutive weekdays
  Interventions: Device: High-frequency repetitive transcranial magnetic stimulation
- Group 3 (Sham Comparator): Sham repetitive transcranial magnetic stimulation: use of a specially fabricated coil that provides no magnetic stimulation but has a similar appearance and creates an auditory artifact that mimics TMS
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Low-frequency repetitive transcranial magnetic stimulation
  Other Names: Nexstim eXimia TMS stimulator with neuronavigation
  Arms: Group 1
Device: High-frequency repetitive transcranial magnetic stimulation
  Other Names: Nexstim eXimia TMS stimulator with neuronavigation
  Arms: Group 2
Device: Sham repetitive transcranial magnetic stimulation
  Arms: Group 3

SUMMARY:
The overall goal of this study is to open up the promising treatment of repetitive transcranial magnetic stimulation (rTMS), which has been shown to be effective against seizures in patients with surface neocortical foci, to a much larger population of patients with mesial temporal lobe epilepsy (MTLE) and other forms of epilepsy with deep foci, who are not currently considered good rTMS candidates.

The investigators hypothesize that rTMS can modulate the hyperexcitable state in patients with deep seizure foci by targeting its usage to accessible cortical partner regions. In this study the investigators aim 1) to map the functional connectivity of the epileptogenic mesial temporal lobe in patients with medically refractory mesial temporal lobe epilepsy; and 2) to perform a randomized controlled assessment of repetitive transcranial magnetic stimulation protocols applied to specific neocortical targets in mesial temporal lobe epilepsy. The methods used in this study will include magnetic resonance imaging (MRI) of the brain, electroencephalography (EEG), and transcranial magnetic stimulation (TMS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mesial temporal lobe epilepsy based on the combination of clinical semiology, neuroimaging findings, and electroencephalogram results.
* At least 1 seizure with loss of awareness per 4-week period, on average, despite the use of antiepileptic drugs

Exclusion Criteria:

* Prior brain surgery or exposure to transcranial magnetic stimulation
* Rapidly progressive brain lesions
* Inability to tolerate MRI or TMS
* Specific MRI or TMS contraindication as set forth in standard protocols of our institution

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-01; Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard S Chang, MD, MMSc, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Low-frequency repetitive transcranial magnetic stimulation: 30-minute sessions of 1-Hz continuous stimulation at 95% resting motor threshold, with one session each day over 10 consecutive weekdays
  Low-frequency repetitive transcranial magnetic stimulation
- Group 2: High-frequency repetitive transcranial magnetic stimulation: 30-minute sessions of 10-Hz continuous stimulation at 110% resting motor threshold, with one session each day over 10 consecutive weekdays
  High-frequency repetitive transcranial magnetic stimulation
- Group 3: Sham repetitive transcranial magnetic stimulation: use of a specially fabricated coil that provides no magnetic stimulation but has a similar appearance and creates an auditory artifact that mimics TMS
  Sham repetitive transcranial magnetic stimulation
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 5 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We were unable to recruit participants for Groups 2 and 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 5 | 0 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 5 |  |  | 5
  >=65 years | 0 |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  |  | 3
  Male | 2 |  |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 5 |  |  | 5
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 1 |  |  | 1
  White | 4 |  |  | 4
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  |  | 5
self-reported seizure frequency [Mean (Standard Deviation); unit: seizure days per 4-week interval] — The baseline measure of the primary outcome will be the self-reported frequency of seizures with loss of awareness, as recorded by participants in written seizure diaries to be provided to the investigators at the end of the 12-week baseline period before intervention. This seizure frequency will be expressed as the number of days on which seizures with loss of awareness occurred per 4-week interval during the baseline period.
  seizure days per 4-week interval | 6.4 (5.4) |  |  | 6.4 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Seizure Frequency
Description: The primary outcome measure will be the self-reported frequency of seizures with loss of awareness, as recorded by participants in written seizure diaries to be provided to investigators at the end of the 12-week assessment period beginning with the initial day of intervention. This seizure frequency will be expressed as the number of days on which seizures with loss of awareness occurred per 4-week interval during the assessment period.
Time Frame: 12 weeks
Population: Group 1 comprised 5 participants. We were unable to recruit participants for Groups 2 and 3.
Measure: Mean (Standard Deviation); unit: seizure days per 4 weeks
Arm/Group | Group 1
Number analyzed (Participants) | 5
seizure days per 4 weeks | 6.4 (5.4)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Group 1
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT02339376/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT02339376/ICF_001.pdf